CLINICAL TRIAL: NCT06954103
Title: Mechanisms And Prognosis of Stroke-Heart Syndrome
Acronym: MAP-SHS
Status: Recruiting | Type: Observational
Sponsor: Chensheng Pan (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Sponsor-Investigator, Chensheng Pan, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: TJ-IRB202502010
Record Dates: First submitted 2025-04-15; First posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-02

CONDITIONS: Stroke; Myocardial Injury; Heart Failure; Acute Coronary Syndromes; Arrhythmia; Sudden Cardiac Death; Takotsubo Syndrome; Heart Rate Variability
Keywords: Stroke-heart syndrome
MeSH Terms: conditions — Stroke; Heart Failure; Acute Coronary Syndrome; Arrhythmias, Cardiac; Death, Sudden, Cardiac; Takotsubo Cardiomyopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma extracted from peripheral blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The incidence of stroke-heart syndrome following acute stroke, which encompasses both acute ischemic stroke and acute intracerebral hemorrhage, is notably high and is strongly associated with increased mortality and poor outcomes in stroke patients. However, the underlying mechanisms remain unclear, and there are currently no effective prevention or treatment strategies. This study aims to elucidate the neuro-humoral mechanisms of stroke-heart syndrome through multimodal imaging and multi-omics blood analysis. Additionally, it seeks to observe the progression of stroke-heart syndrome and its impact on functional outcomes, cognitive abilities, and emotional issues post-stroke. The research is expected to uncover novel blood biomarkers and brain network mechanisms associated with stroke-heart syndrome, providing potential targets and theoretical foundations for pharmacological treatments or physical interventions. Furthermore, it aims to establish a risk early-warning system for major cardiovascular complications post-stroke, enabling early identification, early intervention, and integrated brain-heart management to improve clinical outcomes for stroke patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients admitted within 48 hours of onset, confirmed by CT/MRI as having a stroke (including acute ischemic stroke and hemorrhagic stroke).
2. Moderate-to-severe stroke with NIHSS ≥ 5.

Exclusion Criteria:

1. Previous focal brain injury (such as stroke, brain surgery, traumatic brain injury, etc.).
2. Brain dysfunction caused by other major neurological disorders than stroke (such as brain tumors, epilepsy, Parkinson's disease, etc.).
3. Transient ischemic attack (TIA) and subarachnoid hemorrhage (SAH).
4. History of cardiac diseases (such as coronary heart disease, heart failure, severe arrhythmias, congenital heart disease, cardiac surgery, valvular heart disease, or undiagnosed significant cardiac symptoms).
5. Concomitant systemic diseases such as renal failure (eGFR < 30), autoimmune disorders, severe infections, etc.
6. History of dementia, depression, or other psychiatric disorders.
7. Poor compliance and inability to cooperate with follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be selected from the neurology outpatient clinic, emergency department, and intensive care unit.
Sampling Method: Non-Probability Sample
Enrollment: 658 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
blood high-sensitivity cardiac troponin level | within 48 hours and at 72 hours after stroke onset
  a marker of acute myocardial injury
left ventricular ejection fraction | within 1 week after stroke onset
  measured by transthoracic echocardiography; a marker of ventricular dysfunction and heart failure
blood N-terminal pro-brain natriuretic peptide (NT-proBNP) level | within 1 week after stroke onset
  a marker of ventricular dysfunction and heart failure
functional outcome | 3 months and 1 year after stroke onset.
  measured by modified Rankin scale (mRS), a 7-level ordinal scale (scores 0-6) used to assess global disability after stroke. Higher scores indicate worse functional outcome.
death | 1 month, 3 months and 1 year after stroke onset

SECONDARY OUTCOMES:
post-stroke cognitive impairment | 3 months and 1 year after stroke onset.
  measured by Montreal Cognitive Assessement (MoCA), a widely used screening tool designed to detect mild cognitive impairment and dementia. MoCA score range: 0-30, higher scores indicate better cognitive function.
post-stroke depression | 3 months and 1 year after stroke onset.
  measured by Hamilton depression rating scale (HAMD), a widely used clinician-administered tool for assessing the severity of depression. HAMD score range: 0-52. Higher scores indicate higher depression severity.
post-stroke anxiety | 3 months and 1 year after stroke onset.
  measured by Hamilton anxiety rating scale (HAMA), a clinician-administered tool to assess the severity of anxiety symptoms. HAMA score range: 0-56. Higher scores indicate higher anxiety severity.

CONTACTS AND LOCATIONS:
Overall Officials: Zhou Zhu, MD, PhD, Principal Investigator — Tongji Hospital, Tongji Medical College, Huazhong University of Science and Tech
Locations (1):
- Department of Neurology, Tongji hospital, Tongji medical college, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No